CLINICAL TRIAL: NCT00501787
Title: Tailored Versus Non-tailored Metformin Protocol for Ovulation Induction in Infertile Anovulatory PCOS Patients. A Randomized Controlled Clinical Study
Brief Title: Metformin Administration in Infertile Anovulatory PCOS Patients
Status: Withdrawn | Phase: Phase 4 | Type: Interventional
Sponsor: University Magna Graecia (Other)
Responsible Party: Principal Investigator, Stefano Palomba, Associate Professor, University Magna Graecia
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 05/2006d
Record Dates: First submitted 2007-07-12; First posted 2007-07-16 (Estimated); Last update posted 2013-04-09 (Estimated); Status verified 2013-04

CONDITIONS: Polycystic Ovary Syndrome
Keywords: Anovulation; metformin; PCOS; treatment
MeSH Terms: conditions — Polycystic Ovary Syndrome; Anovulation | interventions — Metformin

ARMS (2):
- Group B (Active Comparator): Non-tailoring
  Interventions: Drug: Metformin
- Group A (Active Comparator): Tailoring
  Interventions: Drug: Metformin

INTERVENTIONS:
Drug: Metformin

SUMMARY:
In a recent prospective study evaluating the efficacy of 1700 mg/day metformin as first-line approach for infertile anovulatory patients with PCOS, we identified predictors for metformin efficacy. Our analysis demonstrated that body mass index (BMI) and insulin resistance were the strongest predictors for both ovulation and pregnancy. In particular, adjusting the data for insulin resistance, a trend in reduced effectiveness was observed with increasing BMI. On the other hand, adjusting the data for BMI, a trend in improved efficacy was detected for higher insulin resistance degrees.

To date, no dose-finding study is currently available in literature evaluating the best dose of metformin to administer. In addition, very few data regarding the best protocol for metformin treatment also are available. However, in order to reduce drug-related side effects incidence due to start-up syndrome, metformin is generally administrated with meals at incremental weekly doses until the maximum dosage ranging from 500 to 2550 mg daily; the doses are reduced if side effects appear. This commonly accepted protocol has not been supported by scientific evidences.

The aim of the present study will be to evaluate in a clinical setting the compliance, the safety and the effectiveness of two schedules for metformin administration in infertile anovulatory PCOS patients.

DETAILED DESCRIPTION:
Infertile anovulatory PCOS eligible patients will be enrolled and randomly allocated to receive tailored (tailored group) or non-tailored metformin treatment (non-tailored group).

Tailored metformin treatment will consist of incremental doses regimen starting from a dosage of 850 mg daily (one tablet daily) with a weekly increase up to 2550 mg daily (three tablets daily). The dosage of metformin will be reduced according to the appearance of serous or affecting compliance drug-related side effects. Conversely, non-tailored metformin treatment consisted of fixed doses regimen of 850 mg twice daily. For both groups, the treatment will be of six months.

All patients eligible will undergo baseline assessment consisting of anthropometric, hormonal, and ultrasonographic evaluations. During the study, the clinical and reproductive outcomes, and the adverse experience will be evaluated in each patient.

Data will be analyzed using the intention-to-treat principle and a P value of 0.05 or less will be considered significant. Continuous variables will be analyzed with the unpaired t test and general linear model for repeated measures analysis with Bonferroni test for the post-hoc analysis as required. For categorical variables, the Pearson chi-square and Fisher's exact tests will be used.

ELIGIBILITY:
Inclusion Criteria:

* Polycystic ovary syndrome (using NIH criteria)
* Anovulatory infertility (using WHO criteria)

Exclusion Criteria:

* Age <18 or >35 years
* Severe obesity (BMI >35)
* Neoplastic, metabolic, hepatic, and cardiovascular disorders or other concurrent medical illnesses
* Hypothyroidism, hyperprolactinemia, Cushing's syndrome, and non-classical congenital adrenal hyperplasia Current or previous (within the last six months) use of oral contraceptives, glucocorticoids, antiandrogens, antidiabetic and anti-obesity drugs or other hormonal drugs
* Previous use of ovulation induction agents
* Intention to start a diet or a specific program of physical activity
* Organic pelvic diseases
* Previous pelvic surgery
* Suspected peritoneal factor infertility
* Tubal or male factor infertility or sub-fertility

Ages: 18 Years to 35 Years | Sex: Female
Age Groups: Adult
Enrollment: 0 (Actual)
Dates: Start 2008-01; Primary Completion 2012-10 (Actual)

PRIMARY OUTCOMES:
Ovulation rate

SECONDARY OUTCOMES:
Adverse events
Adherence rate
Pregnancy rate
Abortion rate
Live-birth rate

CONTACTS AND LOCATIONS:
Overall Officials: Stefano Palomba, MD, Principal Investigator — Department of Obstetrics & Gynecology, University "Magna Graecia" of Catanzaro; Francesco Orio, MD, Principal Investigator — Department of Endocrinology, University "Federico II" of Naples; Achille Tolino, MD, Principal Investigator — Department of Obstetrics & Gynecology, University "Federico II" of Naples
Locations (1):
- Pugliese Hospital, Catanzaro, Catanzaro, CZ, Italy